CLINICAL TRIAL: NCT04979728
Title: HIV Outpatient Monitoring Evaluation Through Self-collection of Dried Blood Spots (HOME-1)
Brief Title: HIV Outpatient Monitoring Evaluation Through Self-collection of Dried Blood Spots
Acronym: HOME-1
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-0382; R01AI170298 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: HIV Treatment; HIV Prevention
Keywords: antivirals; ART; PrEP; long-acting; cabotegravir; rilpivirine; tenofovir; lenacapavir; self-collections; self-collected blood samples; drug concentrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, dried blood samples, capillary blood, plasma, blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Oral Antivirals: Arm 1: People continuing oral (PO) antivirals for HIV treatment or prevention
  Interventions: Other: At Home Self-Collections
- Q8W CAB±RPV Continuation: Arm 2: People continuing Q8W injections of CAB±RPV for HIV treatment or prevention
  Interventions: Other: At Home Self-Collections
- Q8W CAB±RPV Initiation: Arm 3: People initiating Q8W injections of CAB±RPV for HIV treatment or prevention
  Interventions: Other: At Home Self-Collections
- Q4W CAB±RPV Continuation/Initiation: Arm 4: People continuing or initiating Q4W injections of CAB±RPV for HIV treatment or prevention
  Interventions: Other: At Home Self-Collections
- Q26W LEN Continuation/Initiation: Arm 5: People continuing or initiating Q26W injections of LEN for HIV treatment or prevention
  Interventions: Other: At Home Self-Collections

INTERVENTIONS:
Other: At Home Self-Collections — Directly observed at home self-collection of blood samples
  Other Names: Tasso-M20; Tasso+; Mitra; DBS by fingerstick

SUMMARY:
The goal of this observational study is to establish an operational framework for home self-collections of blood samples to be used for antiviral drug concentration measurements.

Participants will continue on their prescribed antiviral(s) for HIV treatment or prevention and followed for up to approximately 1 year. The investigators will compare drug concentrations of antivirals and relevant metabolites/anabolites in clinic-collected and self-collected blood samples.

DETAILED DESCRIPTION:
Up to 150 people receiving care at the UCH-IDGP will be enrolled in the study at a routine clinic visit where a standard of care (SOC) blood collection and/or SOC dose of LA antivirals (e.g., LA IM CAB±RPV) is planned. Once consented, demographic and clinical data will be obtained. Clinical data that will be collected from participant and medical records may include: age, sex at birth and gender identity, race, ethnicity, medication history, duration of current antiviral therapy, hematocrit, CD4+ T-cell count, HIV VL, and self-reported adherence.

The investigators will collect an extra ~5 mL of blood in EDTA by venipuncture for DBS, plasma, whole blood, and blood cells at each clinic-collection visit. At the first clinic-collection visit, participants will be given home self-collection kits and instructed to self-collect samples at various timepoints prior to their next injection (if on LA antivirals), monitored by live video-streaming or time-stamped video. The investigators will go through how to self-collect, handle, and mail the blood samples by self-collecting together in the clinic (in-person training), and participants will be asked about their medical history and medications.

Participants on PO antivirals (e.g., TFV/FTC) may only complete one clinic-collection visit (and one at-home self-collection). At home self-collections and clinic-collections may continue for participants on LA antivirals (e.g., LA IM CAB±RPV) for up to approximately 1 year. All study visits will be linked to SOC visits; there will be no additional visits to the clinic beyond what is already required for SOC:

* If continuing prescribed Q8W injections, up to 7 SOC clinic visits at (approximately) weeks 0, 8, 16, 24, 32, 40, and 48
* If initiating prescribed Q8W injections, up to 7 SOC clinic visits at (approximately) weeks 0, 4, 12, 20, 28, 36, and 44
* If continuing or initiating prescribed Q4W injections, up to 13 SOC clinic visits at (approximately) weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
* If continuing or initiating prescribed Q26W injections, up to 3 SOC clinic visits at (approximately) weeks 0, 26, and 52

Participants will be asked to self-collect samples at home by two or more methods (self-collection kits): fingerstick and spotting onto Whatman 903 protein saver card, and/or use of one or more self-collection devices (e.g., Tasso-M20/Tasso+, Mitra, others). After sample collection, samples/devices will be shipped back to our laboratory in their provided box(es). All samples obtained by self-collection methods/devices are approved for shipping via mail or other carriers in the US. Participants may complete up to 25 at home self-collections (approximately once biweekly for the participants followed longitudinally).

ELIGIBILITY:
Inclusion criteria:

* ≥18 years old
* Receiving one or more antivirals for HIV treatment or prevention. This may include TFV (as TDF or TAF) and FTC (or 3TC)-based, LA (e.g., LA IM CAB±RPV Q4W or Q8W), or other antivirals (those who are transitioning to LA antivirals [e.g., LA IM CAB±RPV Q4W or Q8W] will also be eligible)
* Current patient at the UCH-IDGP clinic
* Able to comply with study procedures, including directly observed self-collection of DBS by fingerstick, Tasso-M20/Tasso+, Mitra, and/or other self-collection methods/devices, and completion of survey

Exclusion criteria:

* Inability to provide informed consent
* Unable or unwilling to comply with directly observed self-collection of DBS (e.g., unavailable or unable to use live video-streaming or time-stamped video recording technology)
* Any uncontrolled medical, social, or mental health issue(s) that, in the opinion of the investigators, could interfere with the study participation or study outcomes (e.g., current incarceration)
* Any medical condition that, in the opinion of the study team, acutely and/or transiently influences the PK of CAB±RPV, including acute kidney injury, hepatic insufficiency, significant drug-drug interactions, active hemolysis or symptomatic hemoglobinopathies, etc. (Note: Given the need for PK data in pregnancy, women who become pregnant while on LA IM CAB±RPV Q4W or Q8W will be allowed to participate in this study, if their clinical provider decides to continue this regimen.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be invited to participate in the HOME-1 study by enrolling a convenience sample of people receiving TFV (as TDF or TAF) and FTC (or 3TC)-based, LA (e.g., LA IM CAB±RPV Q4W or Q8W), or other antivirals for HIV treatment or prevention at the UCH-IDGP. Study visits will only be conducted when blood is to be collected for routine SOC clinical laboratory tests and/or a SOC dose of LA antivirals is to be given.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement of drug concentrations of antivirals and relevant metabolites/anabolites in blood samples | Up to approximately 1 year
  Drug concentrations will be quantified and compared between clinic-collected and at home self-collected samples.

SECONDARY OUTCOMES:
Acceptability of at home self-collection of blood samples | One-time, approximately 1-2 weeks after first clinic-collection visit
  Acceptability will be assessed using the Acceptability of Intervention Measure (AIM). The AIM consists of four questions. For each question, responses range from 1-5, with 1 = completely disagree and 5 = completely agree. The responses to the four questions are then averaged to get an overall acceptability score.
Feasibility of at home self-collection of blood samples | One-time, approximately 1-2 weeks after first clinic-collection visit
  Feasibility will be assessed using the Feasibility of Intervention Measure (FIM). The FIM consists of four questions. For each question, responses range from 1-5, with 1 = completely disagree and 5 = completely agree. The responses to the four questions are then averaged to get an overall feasibility score.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital (UCHealth), Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No